CLINICAL TRIAL: NCT01010100
Title: A Multi-centre, Parallel, Double-blind, Randomised and Placebo Controlled Spanish Study, to Prevent or Delay the Development of Type 2 Diabetes in Subjects With Impaired Glucose Homeostasis Treated With Acarbose in Primary Care (PREDIAP)
Brief Title: Prevent/Delay Development of Type 2 Diabetes in Subjects With Impaired Glucose Homeostasis Treated With Acarbose in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10139; PREDIAP
Record Dates: First submitted 2009-10-26; First posted 2009-11-09 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes Mellitus
Keywords: Metabolic Disease; IGT Impaired Glucose Tolerance
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Glucose Intolerance | interventions — Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acarbose (Glucobay, BAYG5421) — 50 mg TID
  Arms: Arm 1
Drug: Placebo — 50 mg TID
  Arms: Arm 2

SUMMARY:
The purpose of the study is to determine if the administration of small doses of Acarbose can prevent or delay the appearance of Type 2 Diabetes Mellitus in a population of subjects with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 40 and < 75 years old
* Men and women
* Able to give voluntary informed consent
* Existence of one or more of the following risk factors:
* Body Mass Index (BMI) > 27 mg/Kg2
* One or more family members with diabetes determined by anamnesis.
* Personal antecedents of previous blood glucose anomalies (gestational diabetes reverted after the lactation time, before-during surgical stress, fasting glycaemia > 110 mg/dL (6,1 mM) and < 126 mg/dL (7 mM) registered in the Clinical History during the last 3 years, etc.)
* Previous consumption of drugs with hyperglycaemic capacity for a period of 3 months continuously or more than 6 months discontinuously

Exclusion Criteria:

* Type 2 DM
* Pregnancy during the study
* Nursing women
* Major debilitating (e.g. collagen vascular diseases, failure of major organ, psychosis, severe infections, neutropenia, BMI < 20 mg/Kg2)
* Subjects taking a prohibited drug (see protocol)
* Subjects taking drugs that can impair intestinal motility and/or carbohydrate absorption (i.e. cholestyramine, neomycin)
* Recent cardiovascular events (within last 6 months) such as myocardial infarction, cerebrovascular accident, congestive heart failure
* Serum creatinine > 2 mg/Dl
* Fasting triglycerides > 10 mm/L (> 885 mg/dL)
* AST elevation > 2.5 times above the upper limit of normal
* Subjects with hyper/hypothyroidism non compensated
* Subjects with documented gastrointestinal diseases that are likely to be associated with abnormal intestinal motility or altered absorption of nutrients (e.g. gastroparesia, malabsorption syndrome, chronic diarrhoea states, enteropathies, inflammatory bowel diseases, partial intestinal obstruction, large hernias)
* Subjects with any emotional disorder or substance abuse (e.g. severe depression, alcohol or drug abuse)
* Hypersensitivity to Acarbose

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2000-08; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The principal objective was to determine if the administration of small doses of Acarbose could prevent or delay the appearance of Type 2 DM in a population of subjects with impaired glucose homeostasis. | The main criterion for the evaluation of the primary objective was the proportion of diabetic subjects after three years of treatment and another time after three months of wash-out with placebo.

SECONDARY OUTCOMES:
Regression to the normality (NO impaired glucose homeostasis) | Proportion of subjects that had regressed to normality after three years of treatment.
Evolution of the cardiovascular risk markers (microalbuminuria, triglycerides, fasting glycaemia, after overload glycaemia, HbA1c, C-peptide, insulinemia) | Three years and three months.
Evolution of blood pressure | Three years and three months.
Evolution of lipid profile | Three years and three months.
Evolution of anthropometric measurements | Three years and three months. (BMI)
The appearance or progression of cardiovascular events: angina, myocardial infarction, cerebrovascular accident, congestive heart failure, peripheral vascular disease, revascularisation procedure | Time until the appearance or progression of cardiovascular episodes
Delay in the conversion to diabetes mellitus | Time until the confirmation of the diagnosis of Diabetes Mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (20):
- Spain (20):
  - Agost, Alicante
  - Alicante, Alicante
  - Crevillent, Alicante
  - Novelda, Alicante
  - San Vicent del Raspeig, Alicante
  - Terrassa, Barcelona
  - Trobajo del Camino, León
  - Begonte, Lugo
  - Villalba, Lugo
  - Madrid, Madrid
  - Camas, Sevilla
  - Constantí, Tarragona
  - Cornudella, Tarragona
  - el Morell, Tarragona
  - Falset, Tarragona
  - les Borges del Camp, Tarragona
  - Reus, Tarragona
  - Tarragona, Tarragona
  - Tortosa, Tarragona
  - Vinebre, Tarragona